CLINICAL TRIAL: NCT03850886
Title: Evaluation of Efficacy and Safety of Nicotinamide in Non-Alcoholic Fatty Liver Disease Patients
Brief Title: Nicotinamide in Non-Alcoholic Fatty Liver Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rasha Roshdy Ibrahim El-kady, Teaching assisstant at department clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL79
Record Dates: First submitted 2019-01-30; First posted 2019-02-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Niacinamide; Hypoglycemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Niacinamide group (Experimental): Niacinamide oral tablets as Nature's Life 1000 mg tablets once daily for 3 months diabetes management including metformin or Sulphonylurea
  Interventions: Dietary Supplement: Niacinamide Oral Tablet; Drug: Antidiabetic
- Control group (Active Comparator): diabetes management including metformin or Sulphonylurea
  Interventions: Drug: Antidiabetic

INTERVENTIONS:
Dietary Supplement: Niacinamide Oral Tablet — Nature's Life Niacinamide 1000 mg
  Other Names: Nicotinamide; Vitamin B3
  Arms: Niacinamide group
Drug: Antidiabetic — Metformin or Sulphonylurea

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Niacinamide supplementation on clinical outcome of fatty liver patients having type II DM through measurement of the following before and after Niacinamide administration: Liver enzymes, Lipid profie, HOMA-IR, Oxidative stress markers and endothelial dysfunction marker. Fibroscan with CAP will be done at baseline and at the end of the trial. Also, Evaluation of quality of life of patients before and after Niacinamide administration using Chronic Liver Disease questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female outpatients age 18 to 70 years old. 2. The diagnosis of NAFLD will be established according to the appearance of fatty liver on US or elevated liver enzymes (>1.5 times normal level).

Exclusion Criteria:

* 1. History of alcohol abuse (as defined by an average daily consumption of alcohol > 30 g/day in men and > 20 g/day in women).

  2. Cirrhotic patients.
* Fibroscan result > 12Kpa or as
* predicted from FIB 4 score > 3.25

FIB-4 = age (yr) * AST (IU/L)/platelet count (109/L) * ALT1/2 (IU/L) 3. Hyper / hypoparathyroidism. 4. Cancer. 5. Viral hepatitis. 6. Biliary disease. 7. Autoimmune hepatitis 8. Other causes of liver disease (hemochromatosis, Wilson's disease). 9. Participants who took antibiotics, probiotic supplements and/or hepatotoxic medicines (NSAIDs, Amiodarone and methotrexate) within 6 months before the start of the study and during the study.

10. Ascetic patients and congestive heart failure patients will be excluded due to unreliability of Fibroscan results in them.

11. Pregnancy and lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Steatosis using Fibroscan with CAP | 3 months
  using Fibroscan with CAP
Adiponectin mesurement | 3 months
  Endothelial dysfunction

SECONDARY OUTCOMES:
Malondialdehyde | 3 monthes
  Oxidative stress marker
HOMA-IR | 3 months
  Insulin resistance
ALT, AST | 3 months
  Liver enzymes
LDL, cholesterol | 3 months
  Lipid markers

OTHER OUTCOMES:
Chronic Liver Disease Questionnaire | 3 months
  quality of measurement

CONTACTS AND LOCATIONS:
Locations (1):
- AlZahraa hospital, Cairo, Egypt

REFERENCES:
- [Derived] El-Kady RR, Ali AK, El Wakeel LM, Sabri NA, Shawki MA. Nicotinamide supplementation in diabetic nonalcoholic fatty liver disease patients: randomized controlled trial. Ther Adv Chronic Dis. 2022 Feb 23;13:20406223221077958. doi: 10.1177/20406223221077958. eCollection 2022. PMID 35222903